CLINICAL TRIAL: NCT05778357
Title: The Effect of the Covid 19 Pandemic Process on the Neuromotor Developments of 6-24 Month-old Babies: A Cross-sectional Study From Turkey
Brief Title: The Effect of the Covid 19 Pandemic Process on the Neuromotor Developments of 6-24 Month-old Babies
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gökçen Erol, MSc Physiotherapist, Istanbul University - Cerrahpasa
Other Study IDs: GErol
Record Dates: First submitted 2023-03-19; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Development, Infant; Development Delay
Keywords: alberta infant motor scale; denver II developmental screening test; covid-19 pandemic; pediatric rehabilitation
MeSH Terms: conditions — Learning Disabilities; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of neuromotor development of healthy infants: 75 healthy infants were included. Neuromotor development was evaluated with the Denver II Developmental Screening Test and Alberta Infant motor scale.
  Interventions: Other: Group1

INTERVENTIONS:
Other: Group1 — 75 healthy infants were included. Neuromotor development was evaluated with the Denver II Developmental Screening Test and Alberta Infant motor scale.

SUMMARY:
Development; It covers the areas of physical, mental, emotional and social development. Development in one area affects other areas as well. Infancy is the period in which children grow and develop the fastest. Babies need many environmental factors and stimulants in order to have a healthy developmental process. For the Covid 19 pandemic, many restrictions have been made in Turkey to reduce the spread of the epidemic and to maintain social distance between people. It has been suggested that individuals practice their own social isolation. It has also caused babies who spend their time at home during the pandemic process to be deprived of environmental stimuli. In current studies in the literature, it has been reported that the COVID-19 pandemic affects infant and child development significantly and negatively. It has been reported that the risk of delay in children who have experienced the COVID-19 pandemic is especially in the fine motor and communication areas. There is a limited number of studies in the literature on this subject. No study was found in Turkey. The aim of this study is to evaluate the neuromotor development of infants in early childhood (6-24 months) in the Covid-19 pandemic and to reveal the effects of the pandemic process. Denver II Developmental Screening Test was used to evaluate the neuromotor development of healthy infants aged 6-24 months, who applied to the healthy pediatric outpatient clinic of Acıbadem Altunizade Hospital, and Alberta Infant Motor Scale was used to evaluate gross motor functions.

DETAILED DESCRIPTION:
It is an observational study. Purpose of the study: evaluating the neuromotor development of infants in early childhood (6-24 months) in the Covid-19 pandemic and revealing the effects of the pandemic process.

75 healthy infants aged 6-24 months were included.

* Will there be developmental delays in children born in the Covid 19 pandemic?
* In which parameter delay is observed the most.

Denver II Developmental Screenin Test and Alberta Infant Motor Scale were applied to the participants.

ELIGIBILITY:
Inclusion Criteria:

* 75 healthy infants aged 6-24 months were included.

Exclusion Criteria:

* Having a physical/mental/neuromotor/psychological problem
* Not between 6-24 months in the pandemic process
* Presence of a diagnosed disease
* Having a vision problem
* Having a hearing problem

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 75 healthy infants aged 6-24 months were included.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Denver II Developmental Screening Test | baseline
  It is a screening test used in children aged 0-6 years. The test is done in a short time like 5-15 minutes. The person who will administer the Denver II test; must be trained and certified. Standardized test materials are used. The test consists of 4 sections and 134 items. There are personal-social, language, fine motor and gross motor sections. The test result is classified as Normal - Abnormal - Suspicious.
Alberta infant motor scale | baseline
  It is used to observe gross motor functions and evaluate the effectiveness of the intervention in typically developing infants between 0-18 months. The duration of the test is 10 minutes and consists of 58 items. The child's spontaneous movements are evaluated in 4 different positions without touching the child. 1 point is taken for each item that can be done. A table containing the mean and standard deviation for each month is used. The test result is classified as Normal - Abnormal - Suspicious.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.